CLINICAL TRIAL: NCT06108323
Title: Immediate Effects of Mental Practice and Therapeutic Exercise in Mild Smokers: a Randomized Controlled Trial
Brief Title: Immediate Effects of Mental Practice and Therapeutic Exercise in Mild Smokers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Francisco Martínez Arnau, Professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-FIS-2731776-1
Record Dates: First submitted 2023-10-06; First posted 2023-10-31 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Smokers
Keywords: smokers; therapeutic exercise; mental practice; respiratory function
MeSH Terms: conditions — Respiratory Aspiration | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be assigned to one of two study groups by the person conducting the intervention.
  All participants receive mental practice (real or sham) and the exercise program.
  The evaluators are unaware of the assignment at all times.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Action observation plus exercise (Experimental): Therapeutic exercise plus action observation training
  Interventions: Behavioral: Theapeutic exercise plus action observation training
- Sham observation plus exercise (Sham Comparator): Therapeutic exercise plus sham action observation training
  Interventions: Behavioral: Therapeutic exercise plus sham observation training

INTERVENTIONS:
Behavioral: Theapeutic exercise plus action observation training — Participants make an observation of actions related to the training they are going to perform. Subsequently, they perform the therapeutic exercise session.
  Arms: Action observation plus exercise
Behavioral: Therapeutic exercise plus sham observation training — Participants make a sham observation. Subsequently, they perform the therapeutic exercise session.
  Arms: Sham observation plus exercise

SUMMARY:
The goal of this clinical trial is to learn about the effects who would add mental practice based on action observation to a therapeutic exercise program in young mild smokers.

The main question it aims to answer is whether the observation of actions prior to the implementation of a therapeutic exercise session improves the response to it on respiratory, strength and muscle function variables.

Participants will be assigned to one of 2 study groups:

G1) Therapeutic exercise plus action observation training (n=20) G2) Therapeutic exercise plus sham action observation training (n=20)

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Had a pack per year index of <5 (mild smoking index).

Exclusion Criteria:

Those who presented:

* a respiratory pathology,
* cardiac, systematic, or metabolic disease,
* history of recent surgery,
* vertebral fracture,
* or osteoarticular disorders of the spine area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-10-27 (Actual); Primary Completion 2024-04-28 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Respiratory strength | Preintervention and inmediately after the intervention
  Maximal respiratory pressures (in H2O centimeters)

SECONDARY OUTCOMES:
Respiratory function parameters | Preintervention and inmediately after the intervention
  Spirometric parameters (in liters/second)
Physical function | Preintervention and inmediately after the intervention
  5 times sit-to-stand test (in seconds)

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat de Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No